CLINICAL TRIAL: NCT00125268
Title: A Phase III, Double Blind, Randomized, Placebo-controlled Study to Assess the Efficacy of Adjunct Monochromatic Near-infrared Photoenergy (MIRE) in Patients With Painful Axonal Peripheral Neuropathy
Brief Title: Near Infrared Light for the Treatment of Painful Peripheral Neuropathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to enroll enough patients
Sponsor: Mayo Clinic (Other)
Collaborators: Anodyne Therapy, LLC (Industry)
Responsible Party: Matthew Butters, M.D. Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 927-05 00
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Peripheral Neuropathy
Keywords: painful; peripheral; neuropathy; light; therapy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MIRE (Active Comparator): Subjects randomized to this arm will receive treatment with monochromatic near infrared photo energy (MIRE).
  Interventions: Device: MIRE
- Sham (Sham Comparator): Subjects randomized to this arm will receive treatment with the sham device, which is non-active but otherwise identical to the study device.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: MIRE — Monochromatic near infrared photo energy (MIRE). A 30-minute application of MIRE results in a radiant exposure of 43.2 joules per square centimeter (J/cm^2). The design of the flexible pads allows the infrared energy to be delivered perpendicular to and in contact with the involved site. MIRE applied to the skin facilitates the release of a small molecule of the free radical nitric oxide from hemoglobin and other proteins in surrounding tissue. Increased levels of nitric oxide improve the circulation of blood enhancing wound healing and reducing pain.
  Other Names: Anodyne Therapy System
  Arms: MIRE
Device: Sham Device — The sham device is non-active but otherwise identical to the study device.
  Arms: Sham

SUMMARY:
The purpose of this study is to determine if near infrared light therapy is effective in decreasing pain in patients with painful peripheral neuropathy. The hypothesis of the study was that the percentage of subjects with at least 40% improvement in visual analog scale score for pain after 4 weeks of treatment is higher for Monochromatic Near-infrared Photoenergy (MIRE) treatment than for sham treatment.

DETAILED DESCRIPTION:
Pain is a very common symptom, between 65-80%, in patients with peripheral neuropathy. This study is designed to evaluate the effectiveness of monochromatic near infrared photoenergy therapy (MIRE) in the treatment of pain in axonal peripheral neuropathy. This will be compared with a placebo (sham) device.

The MIRE is a FDA approved, drug-free, non-invasive, medical therapeutic device that uses near-infrared light emitting diodes to deliver monochromatic near infrared photoenergy (MIRE) through contact with the skin. The effect of MIRE is believed to increase local blood circulation by dilating vessels and to reduce pain by decreasing local swelling and inflammation. MIRE is also thought to increase local levels of nitric oxide (NO) which may decrease pain levels.

Study subjects will receive treatment with the device or the placebo device 3 times per week for 4 weeks. Response will be measured during and after the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-85; able to give informed consent
* Documented painful, distal peripheral neuropathy of idiopathic cause, or related to impaired glucose tolerance or diabetes mellitus.
* Neuropathy documented by one of the following studies: nerve conduction studies and needle electromyography (EMG); quantitative sensory testing of the foot with Computer Aided Sensory Evaluator (CASE IV); quantitative sudomotor axon reflex test (Quantitative Sweat MeasurementSystem [Q-Sweat]); neurology specialty examination; and neuropathy impairment score (NIS) of less than 25.
* Stable pharmacotherapy for neuropathic pain for at least two weeks.
* Optimal pharmacotherapy has been achieved.
* Subjects cannot be on Cyclooxygenase-2 (COX 2) inhibitors
* Pain Visual Analog Scale (VAS) of greater than or equal to 4/10
* Subject has provided written informed consent
* Not currently using transcutaneous electrical nerve stimulation (TENS)
* Not currently receiving acupuncture

Exclusion Criteria:

* Pregnant or likely to become pregnant
* Current diagnosis of cancer
* Neuropathy impairment score (NIS) of greater than 25.
* Diagnosis of severe neuropathy of known etiology for which specific treatment is available (i.e., acute and chronic inflammatory polyradiculoneuropathies, vasculitis, B 12 deficiency).
* Unstable diabetes mellitus defined as a hemoglobin A1c (HbA1c) greater than 9%, and/or 10% of fasting blood sugars greater than 300 mg/dl for the week prior to enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Butters, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

REFERENCES:
- [Background] Galer BS, Jensen MP. Development and preliminary validation of a pain measure specific to neuropathic pain: the Neuropathic Pain Scale. Neurology. 1997 Feb;48(2):332-8. doi: 10.1212/wnl.48.2.332. PMID 9040716
- [Background] Backonja M, Beydoun A, Edwards KR, Schwartz SL, Fonseca V, Hes M, LaMoreaux L, Garofalo E. Gabapentin for the symptomatic treatment of painful neuropathy in patients with diabetes mellitus: a randomized controlled trial. JAMA. 1998 Dec 2;280(21):1831-6. doi: 10.1001/jama.280.21.1831. PMID 9846777
- [Background] Dyck PJ, Kratz KM, Lehman KA, Karnes JL, Melton LJ 3rd, O'Brien PC, Litchy WJ, Windebank AJ, Smith BE, Low PA, et al. The Rochester Diabetic Neuropathy Study: design, criteria for types of neuropathy, selection bias, and reproducibility of neuropathic tests. Neurology. 1991 Jun;41(6):799-807. doi: 10.1212/wnl.41.6.799. PMID 2046920
- [Background] Holland NR. Idiopathic painful sensory neuropathy. J Clin Neuromuscul Dis. 2001 Jun;2(4):211-20. doi: 10.1097/00131402-200106000-00008. PMID 19078638
- [Background] Kochman AB, Carnegie DH, Burke TJ. Symptomatic reversal of peripheral neuropathy in patients with diabetes. J Am Podiatr Med Assoc. 2002 Mar;92(3):125-30. doi: 10.7547/87507315-92-3-125. PMID 11904323
- [Background] Leonard DR, Farooqi MH, Myers S. Restoration of sensation, reduced pain, and improved balance in subjects with diabetic peripheral neuropathy: a double-blind, randomized, placebo-controlled study with monochromatic near-infrared treatment. Diabetes Care. 2004 Jan;27(1):168-72. doi: 10.2337/diacare.27.1.168. PMID 14693984
- [Background] Mendell JR, Sahenk Z. Clinical practice. Painful sensory neuropathy. N Engl J Med. 2003 Mar 27;348(13):1243-55. doi: 10.1056/NEJMcp022282. No abstract available. PMID 12660389
- [Background] Prendergast JJ, Miranda G, Sanchez M. Improvement of sensory impairment in patients with peripheral neuropathy. Endocr Pract. 2004 Jan-Feb;10(1):24-30. doi: 10.4158/EP.10.1.24. PMID 15251618
- [Background] Koltzenburg M. Painful neuropathies. Curr Opin Neurol. 1998 Oct;11(5):515-21. doi: 10.1097/00019052-199810000-00014. PMID 9848001
- [Background] Wolfe GI, Trivedi JR. Painful peripheral neuropathy and its nonsurgical treatment. Muscle Nerve. 2004 Jul;30(1):3-19. doi: 10.1002/mus.20057. PMID 15221874
- See also: website of company that provided device to be studied — http://www.anodynetherapy.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MIRE | Sham
Started | 16 | 14
Completed | 15 | 13
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MIRE | Sham | Total
Number analyzed (Participants) | 16 | 14 | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 68 (17) | 74 (11) | 71 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects That Have a Greater Than or Equal to Forty Percent Decrease on the Visual Analog Pain Scale at the End of Four Weeks of Treatment
Description: Pain was measured by a 10 cm long Visual Analog Scale (VAS). The VAS does not have any pre-set marks between the extremes. On this scale 0 means no pain and 10 cm means extreme pain. The investigator measures the mark made by the subject in cm and records this for the value of pain.
Time Frame: baseline, 4 weeks
Arm/Group | MIRE | Sham
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Subjects That Have a Forty Percent Reduction of Pain Measured by the Neuropathic Pain Scale at the End of Four Weeks of Treatment
Description: The neuropathic pain scale consists of 10 questions with individual answers rated from 1 to 10, with 0 = no pain to 10 = the most intense pain imaginable. The overall score could range from 0 to 100, with 0 = no pain to 100 = the most intense pain imaginable.
Time Frame: baseline, 4 weeks
Arm/Group | MIRE | Sham
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Subjects That Have an Improvement of Two Points or More on the SF-8 at the End of Four Weeks of Treatment
Description: The SF-8 Health Survey has 8 questions, each question measuring each of the eight domains of health. Scores are calibrated so that 50 is the average score or norm. A lower score indicates poorer health, and a higher score indicates excellent health.
Time Frame: baseline, 4 weeks
Arm/Group | MIRE | Sham
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 4 weeks of the study.
Arm/Group | MIRE | Sham
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/14
Other Adverse Events (participants affected / at risk) | 0/16 | 1/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIRE (N=16) | Sham (N=14)
Carcinoma (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIRE (N=16) | Sham (N=14)
Hypocalcemia (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early because the study was unable to enroll enough patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No